CLINICAL TRIAL: NCT02225938
Title: ICU Recovery: A Multicentre Cohort Study in Critically Ill Patients to Determine Functional Recovery and Quality of Life
Brief Title: ICU Recovery in Australian Patients
Acronym: ICU-RECOVERY
Status: Completed | Type: Observational
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Monash University (Other)
Responsible Party: Sponsor
Other Study IDs: SGS15-0104
Record Dates: First submitted 2014-08-06; First posted 2014-08-26 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2018-08

CONDITIONS: Intensive Care Unit Syndrome
Keywords: Intensive Care; Recovery; Long term outcome; Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intensive care survivors: Patients surviving an admission to an intensive care unit

SUMMARY:
Increasingly patients with critical illness requiring life support in an intensive care unit are surviving their hospital admission. Currently the investigators do not know what effect the ICU admission, and the life support, has on their long-term quality of life and whether they can return to their pre-illness level of function following ICU.

The investigators aim to test telephone follow-up of ICU survivors in assessing function and quality of life six months after ICU admission. Additionally, the investigators will identify if there are factors that lead to poor recovery. The investigators hope this can influence and change current ICU practice to improve recovery and long-term outcomes for patients.

The investigators aim to select a total of 300 patients from ICU, 75 patients from each of the four ICUs. If they survive to hospital discharge, patients and their relatives will receive a telephone questionnaire at 6 months after the ICU admission that aims to assess their long-term outcomes, including physical, cognitive and emotional function, quality of life, and whether they have been able to return to work following ICU.

DETAILED DESCRIPTION:
The ICU Recovery program will measure psychological, functional and cognitive function and quality of life with health economic outcomes in critically ill patients 6 months after ICU admission. The initial pilot study will determine feasibility of the patient outcomes and measurement methods used. The study will consist of patients from three (3) Monash Partners ICUs (2 public and 1 private) as well as The Austin Hospital ICU. 10,000 ICU patients are managed by Monash Partners Academic Health Science Centre (MPAHSC) public and private hospitals each year, of which in the region of 8,500 patients survive. These patients add to the community burden and also influence community and rehabilitation costs. Ultimately, our goal is to establish a national National Health & Medical Research Council (NHMRC) -funded interventional study, led by Monash Partners. Our aim is to improve long-term patient outcomes through: improving sedation practices, delirium prevention, neurocognitive stimulation, early mobilisation, post-ICU follow-up, and functional and psychological rehabilitation. This study is required for the evaluation of hospital and post-ICU rehabilitation practice as there is insufficient evidence to alter current clinical practice.

OBJECTIVES

Primary Aim:

To determine the feasibility of the multi-centre ICU Recovery study using telephone follow-up to assess quality of life, global, psychological, cognitive and physical outcomes at six months following ICU admission.

Secondary Aims

1. To determine the recovery of ICU patients ventilated >24 hours at 6 months after ICU admission
2. To identify risk factors for poor recovery in ICU patients

Tertiary Aims

1. To establish the likely recruitment rate for future studies of long-term outcomes
2. To establish the resource requirements for long term follow-up (including staff, equipment and time taken for survey completion)

ELIGIBILITY:
Inclusion Criteria:

* ICU patients who have been invasively mechanically ventilated for over 24 hours

Exclusion Criteria:

* Patients aged less than 18 years old
* A proven or suspected acute primary brain process that is likely to result in global impairment of conscious level or cognition (e.g. traumatic brain injury, subarachnoid haemorrhage, stroke or hypoxic brain injury after cardiac arrest)
* Second or subsequent admission to ICU during a single hospital admission
* Death is deemed imminent and inevitable
* Participants who do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 critically ill patients who were mechanically ventilated >24 hours in an intensive care unit who have survived to hospital discharge.
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of telephone interview | At completion of telephone interview, expected average of 6 months
  Determine feasibility of using a telephone interview to ascertain the functional recovery and quality of life and critically ill ICU survivors.

SECONDARY OUTCOMES:
Health related quality of life | At telephone interview, conducted at an expected average of 6 months following discharge from the Intensive Care Unit
  Health related quality of life (HRQOL) measured with EuroQol five dimensions questionnaire (EQ-5D) before ICU (retrospective survey) and at 6 months (prospective survey)

OTHER OUTCOMES:
Pre-ICU function | At telephone interview, conducted at an expected average of 6 months following discharge from the Intensive Care Unit
  Pre-ICU function measured with EuroQol five dimensions questionnaire (EQ-5D) and work details
Global function | At telephone interview, conducted at an expected average of 6 months following discharge from the Intensive Care Unit
  Global function at 6 months, assessed with World Health Organization Disability Assessment Schedule (WHODAS)
Physical activity | At telephone interview, conducted at an expected average of 6 months following discharge from the Intensive Care Unit
  Physical activity at 6 months, assessed with International Physical Activity Questionnaire (IPAQ).
Cognitive function | At telephone interview, conducted at an expected average of 6 months following discharge from the Intensive Care Unit
  Cognitive function at 6 months, assessed with Telephone Interview for Cognitive Status (TICS).
Anxiety and depression | At telephone interview, conducted at an expected average of 6 months following discharge from the Intensive Care Unit
  Anxiety and depression at 6 months will be assessed with the Hospital Anxiety and Depression Scale (HADS) and the Impact of Event Scale (IES-R)
Return to work | At telephone interview, conducted at an expected average of 6 months following discharge from the Intensive Care Unit
  Return to work at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carol Hodgson, PhD MRes, Principal Investigator — ANZIC-RC
Locations (5):
- Australia (5):
  - Monash Medical Centre, Clayton, Victoria
  - The Austin Hospital, Heidelberg, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Epworth Hospital, Richmond, Victoria

REFERENCES:
- [Derived] Hodgson CL, Udy AA, Bailey M, Barrett J, Bellomo R, Bucknall T, Gabbe BJ, Higgins AM, Iwashyna TJ, Hunt-Smith J, Murray LJ, Myles PS, Ponsford J, Pilcher D, Walker C, Young M, Cooper DJ. The impact of disability in survivors of critical illness. Intensive Care Med. 2017 Jul;43(7):992-1001. doi: 10.1007/s00134-017-4830-0. Epub 2017 May 22. PMID 28534110